CLINICAL TRIAL: NCT00580346
Title: Dynamic Laryngotracheal Separation for Aspiration. Prevention of Silent Aspiration Pneumonia During Swallowing by an Implanted Stimulator
Brief Title: Dynamic Laryngotracheal Separation for Aspiration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 01-01-02; NIH DC-006703-01; IDE G980179
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Aspiration Pneumonia
Keywords: Aspiration pneumonia; Implanted laryngeal stimulator; Vocal cord closure; Modified barium swallow
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental)
  Interventions: Device: Placement of laryngeal implant

INTERVENTIONS:
Device: Placement of laryngeal implant — Placement of stimulator over anterior chest wall, and electrodes around recurrent laryngeal nerve, and tunneling leads between both
  Other Names: Modified Finetech Vocare Bladder stimulator; Huntington perineural electrodes

SUMMARY:
People who aspirate after neurologic insults such as stroke often develop fatal pneumonia. This study examines the effects of dynamic vocal cord closure on swallowing. Implants placed over the chest wall are connected to electrodes placed around the nerve that closes the vocal cords. The patient triggers closure by flipping the switch of a coil taped over the skin covering the internal stimulator. Vocal cord motion is verified by videotaping through an endoscope, and the status of swallowing is documented radiologically by a modified barium swallow.

DETAILED DESCRIPTION:
Data pending

ELIGIBILITY:
Inclusion Criteria:

* Aspiration pneumonia after neurological insults (e.g. stroke)
* Ability to understand the purpose of the research
* Appropriate hand motor control
* Inability to improve under standard treatments (speech-language pathologists)
* Acceptance of a tracheostomy

Exclusion Criteria:

* Lack of understanding the research
* Poor hand motor coordination
* Uncontrolled seizures
* Pregnancy
* Refusal to accept a tracheostomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Videotaping vocal cords and modified barium swallows | several months

SECONDARY OUTCOMES:
Tolerance of implanted device | immediate to several years
comfort in swallowing | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Broniatowski, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Health System, Cleveland, Ohio, United States

REFERENCES:
- [Background] Broniatowski M, Grundfest-Broniatowski S, Tyler DJ, Scolieri P, Abbass F, Tucker HM, Brodsky S. Dynamic laryngotracheal closure for aspiration: a preliminary report. Laryngoscope. 2001 Nov;111(11 Pt 1):2032-40. doi: 10.1097/00005537-200111000-00031. PMID 11801992